CLINICAL TRIAL: NCT01710111
Title: Evaluating Modes of Influenza Transmission Using a Human Challenge Model
Brief Title: Evaluating Modes of Influenza Transmission
Acronym: EMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Retroscreen Virology Ltd. (Industry); Wake Forest University Health Sciences (Other); University of Maryland (Other); University of Leeds (Other); Building Services Research and Information Association (BSRIA) (Unknown); University College, London (Other); Mount Sinai Hospital, New York (Other); Imperial College London (Other); University of Glasgow (Other); Sydney Children's Hospitals Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12074
Record Dates: First submitted 2012-10-09; First posted 2012-10-18 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Influenza, Human
Keywords: Human challenge model; Quarantine study; Influenza virus; Modes of transmission; Droplet spray; Droplet nuclei; Secondary attack rate; Face shield; Hand hygiene; Fomites; Environmental deposition; Environmental dispersion
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Recipients Face Shield (Experimental): Face shield and repeat hand hygiene measures
  Interventions: Device: Intervention Recipients Face Shield
- Control Recipients (No Intervention): No face shield and no repeat hand hygiene measures

INTERVENTIONS:
Device: Intervention Recipients Face Shield — Face shield and repeat hand hygiene measures
  Arms: Intervention Recipients Face Shield

SUMMARY:
The ways in which influenza is transmitted between people are uncertain; for example, we do not know if large droplets or fine particles (aerosols) matter most; both are produced by coughing and sneezing. This means we cannot say what precautions work best in real life. Improving our understanding is vital to allow the development of guidelines and policies to help reduce the transmission of both pandemic and seasonal flu.

The aim of this study is to explore how influenza is spread, specifically by looking at the importance of spread via small particles (aerosols/droplet nuclei) that are carried in respiratory sprays e.g. produced by coughing and sneezing.

The primary objective of this study is:

To estimate the contribution of aerosols/droplet nuclei to influenza transmission by determining the secondary attack rate (SAR) of influenza in Recipients randomised to a control arm (no intervention - allowing all modes of transmission) compared to Recipients randomised to an intervention arm (face shield and hand hygiene - allowing only transmission by aerosols/droplet nuclei) when both groups of Recipients are exposed to Donor volunteers infected with influenza via intranasal drops.

The hypothesis is that:

The SAR will be lower in Recipients exposed only to aerosols/droplet nuclei (intervention arm) compared to those exposed to all modes of transmission (the control arm): aerosols/droplet nuclei, droplet spray (larger respiratory droplets) and transmission through contact.

DETAILED DESCRIPTION:
The study will take place in a quarantine facility. Some volunteers (Donors) will be infected with the influenza virus via droplets into the nose. Other volunteers (Recipients) will then be exposed to them by occupying the same room (in the day time) and taking part in certain activities e.g. playing card games. Some of the Recipients will wear face shields and clean their hands regularly during the times they are with the Donors. The wearing of face shields together with good hand hygiene should reduce the spread of infection through large respiratory droplets and contact with contaminated surfaces but will not prevent infection that occurs through aerosols in the air. Use of symptom diaries and diagnostic tests for influenza will allow the presence of subsequent illness to be identified. Volunteers will be required to participate in the quarantine facility for up to approximately 13 days (typically 9 for Donors and 13 days for Recipients), plus study screening clinics and followup.

Additionally, during the study, environmental sampling will be performed looking for the presence of influenza virus. Air sampling and swabbing of surfaces and objects may provide information enabling us to better understand the routes of transmission.

ELIGIBILITY:
Inclusion Criteria:

* Body Weight: A total body weight ≥50 kg and a Body mass index (BMI) >18 (if BMI is >32, a body fat percentage within WHO and NIH range for gender and age. BMI [kg/m2] = Body weight [kg] ÷ Height2 [m2]
* Contraception: Nonsterilised males must agree to refrain from fathering a child from the point of entering quarantine until the Day 28 follow up visit. Use of one effective form of contraception is acceptable. Sexually active females of childbearing potential must agree to use 2 effective methods of avoiding pregnancy that are deemed to be effective from the point of entry into the quarantine unit until the Day 28 follow up visit. Acceptable forms of effective contraception include:

  1. Established use of oral, injected or implanted hormonal methods of contraception.
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
  3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
  4. Male sterilisation (with the appropriate postvasectomy documentation of the absence of sperm in the ejaculate). [For female subjects on the study, the vasectomised male partner should be the sole partner for that subject].
  5. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].
* Informed Consent: An informed consent document signed and dated by the subject and investigator
* Serosuitability: Serosuitable for challenge virus

Exclusion Criteria:

* Smoking: Significant history of any tobacco use at any time (≥ total 10 pack year history, eg. one pack a day for 10 yrs)
* Pregnancy/Lactation: Subjects who are pregnant or nursing, or who have a positive pregnancy test at any point in study
* Previous Medical History: Presence of significant acute or chronic, uncontrolled medical illness, that in the view of Investigator(s)is associated with increased risk of complications of respiratory viral illness
* Pulmonary Function: Abnormal pulmonary function in the opinion of the investigator evidenced by clinically significant abnormalities in spirometry
* Immune: History or evidence of autoimmune disease or known impaired immune responsiveness (of any cause)
* Asthma: History of asthma, COPD, pulmonary hypertension, reactive airway disease, or any chronic lung condition of any aetiology.History of childhood asthma until and including the age of 12 is acceptable.
* HIV & Hepatitis: Positive HIV, hepatitis B (HBV), or hepatitis C (HCV) antibody screen.
* Anatomic abnormalites of nasopharynx:Significant abnormality altering anatomy of nose or nasopharynx
* Epistaxis: Clinically significant history of epistaxis
* Nasal Surgery: Any nasal or sinus surgery within 6 months of inoculation
* Fainting: Recent (within the last 3 years of the screening visit) and/or recurrent history of clinically significant autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, etc)
* Lab Test/ECG: Laboratory test or ECG which is abnormal and deemed by investigator(s) to be clinically significant.
* Drugs of abuse etc: Confirmed Positive test for class A drugs or alcohol that cannot be satisfactorily explained
* Venous Access: Venous access deemed inadequate for phlebotomy (and IV infusion) demands of study
* Hayfever: Subjects symptomatic with hayfever on admission or prior to inoculation.
* Allergies: Any known allergies to excipients in challenge virus inoculum
* Healthcare workers: Health care workers (including doctors, nurses, medical students and allied healthcare professionals) anticipated to have patient contact within two weeks of viral challenge. Healthcare workers should not work with patients until 14 days after challenge or until symptoms are fully resolved (whichever is longer). In particular, health care workers who work in units housing, elderly, disabled or severely immunocompromised patients (e.g. bone marrow transplant units) will be excluded.
* Household members: Presence of household member or close contact (for an additional 2 weeks after discharge from the isolation facility) who is:

  1. less than 3 years of age
  2. any person with any known immunodeficiency
  3. any person receiving immunosuppressant medications
  4. any person undergoing or soon to undergo cancer chemotherapy within 28 days of viral inoculation
  5. any person with diagnosed emphysema or chronic obstructive pulmonary disease (COPD), is elderly residing in a nursing home, or with severe lung disease or medical condition that may include but not exclusive to conditions listed (detailed in protocol); or
  6. any person who has received a transplant (bone marrow or solid organ)
* Travel: Intending to travel within next 3 months (to countries for which travel vaccinations are recommended).
* Employers: Those employed or immediate relatives of those employed at RVL or staff/ students working directly for any unit in which CI works.
* Blood loss/receipt: Receipt of blood or blood products, or loss (including blood donations) of 450 mL or more of blood, during the 3 months prior to inoculations.
* Use of nasal congestion products - acute/chronic: Acute use i.e. within 7 days prior to viral challenge of any medication or other product (prescription or OTC), for symptoms of hayfever, rhinitis, nasal congestion or respiratory tract infection.
* Other IMP or virus challenges: Receipt of any investigational drug within 3 months prior inoculation. Receipt of more than 4 investigational drugs within the previous 12 months. Prior participation in a clinical trial with same strain of respiratory virus. Participation in other respiratory virus challenge within 1 year prior to challenge
* Chemotherapy: Receipt of systemic glucocorticoids, antiviral drugs, and immunoglobulin's (Igs) or other cytotoxic or immunosuppressive drug within 6 months prior to dosing. Receipt of any systemic chemotherapy agent at any time.
* Current or recent respiratory infection: Presence of significant respiratory symptoms on day of challenge or between admission for challenge and challenge with/exposure to virus. History suggestive of respiratory infection within 14 days prior to admission for challenge exposure.
* General screening: Any other finding in medical interview, physical exam, or screening investigations that, in the opinion of the investigator, GP or sponsor, deem subject unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference in Secondary Attack Rate (SAR) | Day -2 to day 28(±3)
  The primary endpoint is the difference in SAR of influenza in Recipients randomised to an intervention arm (face shield and hand hygiene -droplet nuclei transmission only) compared to Recipients randomised to a control arm (no intervention - all modes of transmission).

SECONDARY OUTCOMES:
Viral parameters of infection and association with infection transmission. | Day 1 to day 10
  To evaluate and compare the incidence, duration and quantity of human virus shedding.
  To explore and compare the association of the incidence (infection rate as well as daily incidence), duration and quantity of virus shedding in Donors, with transmission to Recipients.
Clinical parameters of infection and association with infection transmission. | Day 1 to day 10
  To explore the association and severity of self-reported influenza symptoms and pyrexia between Recipient groups (intervention vs. no intervention), both cumulatively and by individual symptom type.
  To explore the association of self-reported influenza symptoms in Donors, with transmission to Recipients, both cumulatively and by individual symptom type.
Environmental disposition of virus during infection. | Day 1 to day 10
  To determine the environmental dispersion and deposition of the virus (fomites and air) in Exposure rooms and the relationship between (a) virological findings and environmental deposition, (b) symptom scores and environmental deposition, and (c) environmental deposition and SAR in Recipients.
  To characterize the exhaled breath particle sizes and aerosolized virus copy numbers expelled by influenza inoculated and influenza exposed volunteers.
Safety of experimental infection in both challenged and exposed volunteers. | Day 1 to day 28(±3)
  * Incidence, severity, and relationship of adverse events to challenge virus and/or study procedures.
  * Changes in safety laboratory tests, vital signs and clinical tests (electrocardiogram [ECG], spirometry) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Nguyen-Van-Tam, BM, BS, DM, Principal Investigator — University of Nottingham
Locations (1):
- Retroscreen Virology Ltd, London, United Kingdom

REFERENCES:
- [Derived] Bueno de Mesquita PJ, Noakes CJ, Milton DK. Quantitative aerobiologic analysis of an influenza human challenge-transmission trial. Indoor Air. 2020 Nov;30(6):1189-1198. doi: 10.1111/ina.12701. Epub 2020 Jun 15. PMID 32542890